CLINICAL TRIAL: NCT01813955
Title: PDE Inhibitors Effect on Cognitive Deficits Associated to Schizophrenia
Brief Title: Phosphodiesterase (PDE) Inhibitors Effect on Cognitive Deficits Associated to Schizophrenia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Patient recruitment insufficient
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Birte Glenthoj, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Papaverine schizophrenia
Record Dates: First submitted 2011-09-19; First posted 2013-03-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Cognitive Deficits
Keywords: phosphodiesterase inhibitor; Psychophysiology; Cognition; Schizophrenia; Papaverine
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Papaverine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Papaverine (Experimental): Patients will receive either Papaverine or placebo added to their current medical treatment. Then after one week, they will receive the other treatment (if it was placebo first, then it will be papaverine; if it was papaverine first, then it will be placebo)
  Interventions: Drug: Papaverine or placebo

INTERVENTIONS:
Drug: Papaverine or placebo — Papaverine delayed release (depot capsule, 300 mg, orally, one single dosage per subject) or placebo
  Other Names: Papaverine

SUMMARY:
Phosphodiesterase (PDE) inhibitors represent a new group of potential antipsychotic compounds currently under development. One of these is papaverine, an inhibitor of the PDE 10 family. The class of PDE10 inhibitors have been reported as possible candidates in the treatment of schizophrenia, and may prove an attractive antipsychotic alternative due to the many side-effects of the currently available antipsychotics. It has been proposed from preclinical studies that PDE10 inhibitors have the potential to reduce cognitive deficits in schizophrenia and these findings need to be confirmed in a human population, in view of the fact that no other currently registered drug posses these unique properties.

The currently proposed project is designed to investigate whether the PDE10 inhibitor Papaverine indeed have the capacity to reduce cognitive deficits in schizophrenia patients. In order to accomplish this effect, Papaverine will be investigated in schizophrenia, with regards to symptomatology, hemodynamic, neurocognition and early information-processing.

DETAILED DESCRIPTION:
The study has a double blind, balanced crossover design. Randomized, half of the subjects will be given Papaverine (PDE10 inhibitor, 300 mg orally) in the first session followed by placebo in the second, and the other half will be treated in the reverse order. There is a minimum of one month between the two test-sessions. After each of the two treatments, the subjects will be tested with both a psychophysiological (the Copenhagen Psychophysiological Test-Battery) and neuropsychological test-battery (tests from the Cambridge Neuropsychological Test Automated Battery, or "CANTAB"). The project has three phases: In the first phase 10 healthy subjects will be included to determine the kinetics of Papaverine-contained release capsules ; in the second phase 30 schizophrenia patients and 30 healthy subjects will be included to determine the impact on cognitive and sensory gating related deficits; Finally 10 Healthy subjects will be included to determine the effect of Papaverine on hemodynamical parameters by the means magnetic resonance scannings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Schizophrenia (WHO ICD 10)
* Treatment stable (no regulation in medicine for 6 weeks prior)
* Mono antipsychotic treatment
* No regular Antidepressants (PN accepted)
* No regular Benzodiazepines (PN accepted)

Exclusion Criteria:

* Dependence syndrome
* Severe physical illness
* MRI incompatible, non removable objects above shoulders

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
psychophysiology | 1 hour after intake of capsule with papaverine or placebo
  Prepulse inhibition of the startle reflex, Mismatch negativity, P300 amplitude

SECONDARY OUTCOMES:
Hemodynamic changes | 1 hour after intake of capsule with papaverine or placebo
  Changes in Hemodynamics, as observed by MR techniques

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthøj, Professor, Study Director — University of Copenhagen; Mikkel E Sørensen, PHD student, Principal Investigator — University of Copenhagen; Bob Oranje, PHD, Study Director — Center for Neuropsychiatric Schizophrenia Research
Locations (1):
- Glostrup psychiatric center, Glostrup Municipality, Denmark